Nothing herein is to be disclosed in any way without the prior expressed written permission of W. L. Gore & Associates, Inc.

# Evaluation of the GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis in the Treatment of Thoracoabdominal and Pararenal Aortic Aneurysms

Protocol Number: AAA 17-01

24-Mar-2023

W. L. Gore & Associates, Inc. Medical Products Division

# **PROTOCOL SUMMARY**

| Study Title | Evaluation of the GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis in the Treatment of Thoracoabdominal and Pararenal Aortic Aneurysms |
|---|---|
| Protocol Number | AAA 17-01 |
| IDE Number | G150071 |
| Sponsor | W. L. Gore & Associates, Inc. Telephone: 800-437-8181 |
| Study Design | Prospective, non-randomized, multicenter study with two independent arms: • Primary Study Arm – TAAA requiring only TAMBE System. Hypothesis-driven analysis. • Secondary Study Arm – TAAA requiring TAMBE System and CTAG Device(s). Non-hypothesis-driven analysis. |
| Study Objective | Assess the safety and effectiveness of the TAMBE Device in the treatment of thoracoabdominal and pararenal aortic aneurysms |
| Co-Primary Study<br>Endpoints | Uncomplicated Technical Success / Procedural Safety Co-Primary Endpoint A composite of the following events: • Device Technical Success at the time of the index endovascular procedure • Procedural Safety events within 30 days of index procedure: Clinically Significant Reintervention / Lesion-Related Mortality Co-Primary Endpoint (12 months post-treatment) • Clinically Significant Reintervention (using protocol definition) • Lesion-Related Mortality |
| Subject Population | Subjects with thoracoabdominal or pararenal aortic aneurysms requiring treatment Primary Study Arm: Adapted Crawford Type IV TAAA and Pararenal aneurysms (n= 102) |

| | Secondary Study Arm: Adapted Crawford Type I-III (n= 20 - 100) Continued Access (Primary Study Arm): Adapted Crawford Type IV TAAA and Pararenal Aneurysms (n=up to 65) |
|---|---|
| Number of Implanted<br>Subjects | Minimum: 122 implanted subjects, Maximum: 202 implanted subjects with up to 65 additional subjects implanted in Continued Access (Primary Study arm). |
| Number of Sites | Up to 45 sites in the United States and Europe |
| Coordination PI | |
| Brief Inclusion Criteria | <ul> <li>Aortic aneurysm involving the visceral vessels requiring treatment defined as at least one of the following: <ul> <li>Fusiform aneurysm diameter ≥ 5 cm</li> <li>Saccular aneurysm (no diameter requirement)</li> <li>Rapid aneurysm growth (≥ 5 mm in one year)</li> </ul> </li> <li>An Informed Consent Form signed by Subject or legal representative</li> <li>Appropriate aortic anatomy to receive the TAMBE Device defined as all of the following: <ul> <li>For the TAMBE Aortic Component, proximal aortic landing zone diameters between 22 -34 mm</li> <li>Proximal seal zone ≥ 20 mm in length</li> </ul> </li> </ul> |
| Brief Exclusion Criteria | <ul> <li>Prior open, aortic surgery of the ascending aorta or aortic arch</li> <li>Myocardial infarction or stroke within 1 year of treatment (staged or index procedure)</li> <li>Previous instance of Heparin Induced Thrombocytopenia type 2 (HIT-2) or known hypersensitivity to heparin</li> <li>Renal insufficiency (creatinine value &gt; 1.8 mg/dL, GFR &lt; 30, or patient undergoing dialysis)</li> </ul> |
| Expected Time to<br>Complete Enrollment | Primary Study Arm Subject Accrual: 27-32 months Follow-up – 5 years from last subject enrollment |
| Brief Schedule of<br>Events | Screening Pre-Treatment Treatment Discharge Follow-up (30 day, 3, 6, 12 months and annually thru 5 years) |

# STUDY and VENDOR INFORMATION

| 41 Jan | VENDOR INFORMATION |
|---|---|
| S | Study Information |
| Study Contact Information | General e-mail: Study manager information Emergency Contact Located in the study Regulatory Binder |
| Study Financing | Financed by W. L. Gore & Associates, Inc. |
| Data Monitoring Committees (Gore-coordinated) | Clinical Events Committee (CEC) Data Safety Monitoring Board (DSMB) |
| Emergency and Compassionate Use | Supported, with conditions |
| Reimbursement Information | Reference the Claims Binder |
| Study Roster | List of sites (addresses, principal investigator, emergency contact information) Located in the study Regulatory Binder |
| Ve | endor Information |

Evaluation of the GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis in the Treatment of Thoracoabdominal and Pararenal Aortic Aneurysms

# **Statistical Analysis Plan**

Study Acronym / Protocol #: AAA 17-01

# **Table of Contents**

| 1. | Intro | duction | | 1 |
|---|---|---|---|---|
| | 1.1 | Study | Success | 1 |
| 2. | Study | / Design | Overview | 1 |
| | 2.1 | Object | tives | 2 |
| | | 2.1.1 | Primary Objective(s) | 2 |
| | | 2.1.2 | Secondary Objective(s) | 2 |
| | 2.2 | Desig | n Summary | 2 |
| | 2.3 | Study | Endpoints | |
| | | 2.3.1 | Primary Endpoint(s) | |
| | 2.4 | | Secondary Endpoint(s) | |
| | 2.4 | | ical Hypotheses | |
| | 2.5 | | le Size Assumptions | |
| • | 2.6 | | le Size Calculations | |
| 3. | | • | ent Arms | |
| | 3.1 | | ırms | |
| | 3.2 | | ol Arm(s) | |
| 4. | | • | ollection | |
| | 4.1 | • | Collection Intervals | |
| | 4.2 | | -up Visit Windows | |
| | 4.3 | | and Safety Monitoring Board | |
| | 4.4 | | al Event Committee | |
| | 4.5 | | nrollment Restrictions | |
| | 4.6 | Core L | _ab | 12 |
| | 4.7 | Handli | ng of Missing Dates | 12 |
| 5. | Statis | stical Ana | alyses | 13 |
| | 5.1 | Analys | sis Populations | 13 |
| | 5.2 | Endpo | int Variables | 13 |
| | 5.3 | Timing | g of Analyses | 13 |
| | 5.4 | Statist | ical Analysis of Endpoints | 14 |
| | | 5.4.1 | Uncomplicated Technical Success / Procedural Safety Endpoint Events | 14 |
| | | 5.4.2 | Clinically Significant Reintervention / Lesion Related Mortality Events Endp | |
| | 5.5 | Adver | Eventsse Events | |
| | 5.6 | | onal Analyses | |
| | 0.0 | 5.6.1 | Reduced Alpha Analysis | |
| | | 0.0.1 | | |

# Statistical Analysis Plan

| | | 5.6.2 | Analysis by Potential Confoundi | ng Factors | 15 |
|---|---|---|---|---|---|
| | | | 5.6.2.1 Analysis by Aneurysm 7 | <sup>-</sup> ype | 15 |
| | | | 5.6.2.2 Analysis by Aneurysm S | Size | 15 |
| | | | 5.6.2.3 Analysis of Enrolled but | not Implanted Subjects | 15 |
| | | | 5.6.2.4 Endpoint Analysis by Se | xx | 16 |
| | | | 5.6.2.5 Attrition Sensitivity Anal | yses | 16 |
| | | | 5.6.2.6 Site Pooling | | 16 |
| | | | 5.6.2.7 Analysis of Missing Data | a | 16 |
| | | | 5.6.2.8 Rationale of Number of | Procedures by a Single User | 17 |
| 6. | Interin | n Analys | es and Safety Monitoring Analys | es (if applicable) | 17 |
| 7. | Analys | sis Spec | ications | | 17 |
| | 7.1 | SAS A | alysis Dataset Specifications | | 17 |
| | 7.2 | Statist | al Output Specifications | | 17 |
| | 7.3 | Verific | tion Level for Statistical Output | | 17 |
| 8. | Data 9 | Sets, Ta | les, Figures, and Listings | | 18 |
| | 8.1 | Analys | Tables | | 18 |
| | 8.2 | Analys | Listings | | 18 |
| | 8.3 | Analys | Figures | | 19 |
| 9. | Refere | ences | | | 19 |
| 10 | Povici | on Hict | N. | | 10 |

#### 1. Introduction

This Statistical Analysis Plan (SAP) describes the statistical analyses planned to address the objectives of the AAA 17-01 clinical study. This SAP summarizes the analyses that will be performed to determine the safety and effectiveness of the Thoracoabdominal Branch Endoprosthesis (TAMBE) Device when used for endovascular repair of thoracoabdominal and pararenal aortic aneurysms in subjects with appropriate anatomy. This SAP outlines tables, figures, and listings that are included in reports for the AAA 17-01 clinical study.

## 1.1 Study Success

Study success will be defined as rejecting the null hypotheses from both the Uncomplicated Technical Success Endpoint and the Clinically Significant Reintervention end points.

#### 2. Study Design Overview

This will be a prospective, non-randomized, two-armed, multicenter study conducted at up to forty-five (45) Clinical Investigative Sites (referred to as "sites" in the remainder of this document) in the United States and Europe. A minimum of 122 subjects, up to a potential maximum of 202 subjects, will be implanted with the TAMBE Device across two independent study arms as described below.

- Primary Study Arm Hypothesis-driven analysis, Thoracoabdominal aneurysms (TAAAs) which
  are anatomically suitable for treatment with the TAMBE Device and do not require proximal
  extension with a CTAG Device (N=102). This arm will be limited to pararenal aortic aneurysm and
  adapted Crawford Type IV TAAAs.
- Secondary Study Arm Non hypothesis-driven analysis, TAAAs which are anatomically suitable
  for treatment with the TAMBE Device and would require proximal extension with CTAG Device(s).
  This arm will include adapted Crawford Type I-III TAAAs. (N=20-100 Subjects)

Up to 65 additional subjects may be implanted in the Continued Access Phase under the Primary Study Arm only. All sites will be allowed to enroll in the Continued Access Phase, and all sites and subjects will be treated and followed in the same manner as the Core Clinical Investigation.

- The reduced profile VBX Device cohort (a subset of the Continued Access phase) will follow
  the TAMBE protocol: all primary, secondary, and other endpoints will be collected for these
  subjects as per protocol in the same manner as for the other cohorts. The Target Vessel
  Technical Success of the reduced profile VBX Device for each vessel will also be assessed.
- To assess the compatibility of reduced profile VBX Device as a side branch component in conjunction with the TAMBE Aortic Component (AC), the following endpoints will be summarized at a subject level:
- Uncomplicated Technical Success at Index Procedure
- Procedural Safety data through 30-day follow-up
- Summary of AEs through 30-day follow-up including Type Ic and IIIc Endoleaks



## 2.1 Objectives

## 2.1.1 Primary Objective(s)

The primary objective of the study is to determine whether the GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis is safe and effective in the treatment of thoracoabdominal and pararenal aortic aneurysms.

The study will utilize separate, independent hypothesis-driven analyses in order to make this determination in the study's target population of pararenal aortic aneurysm subjects and adapted Crawford Type IV thoracoabdominal aneurysm subjects.

Gore recognizes that the TAMBE Device, in combination with proximal CTAG Device extension, may have applicability to Crawford Type I-III thoracoabdominal aneurysm subjects. Hypothesis-driven assessments will not be performed in this secondary study arm population with device performance characterized for potential future applications.

#### 2.1.2 Secondary Objective(s)

There are no Secondary Objectives specified for this study.

## 2.2 Design Summary

AAA 17-01 is a prospective, non-randomized, multi-center trial that will compare the Uncomplicated Technical Success / Procedural Safety and Clinically Significant Reintervention / Lesion Related Mortality co-primary endpoints to pre-specified performance goals. A minimum of 122 subjects and a maximum of 202 subjects will be enrolled and implanted across both sub-groups; 102 Subjects within the Primary Study Arm and between 20 and 100 Subjects within the Secondary Study Arm, with a minimum requirement of 20 combined adapted Crawford Type I and Type II aneurysms. Subjects will be evaluated through hospital discharge and return for follow-up visits at one (1), three (3), six (6), 12, 24, 36, 48 and 60 months. This is a confirmatory study.

## 2.3 Study Endpoints

## 2.3.1 Primary Endpoint(s)

There are two Co-Primary Endpoints used in this study: Uncomplicated Technical Success / Procedural Safety and Clinically Significant Reintervention / Lesion Related Mortality. A hypothesis test will be conducted on each Co-Primary Endpoint.

 Uncomplicated Technical Success / Procedural Safety Co-Primary Endpoint (evaluated through 30 days post procedure)

**Table 1** displays the components for the Uncomplicated Technical Success Primary Endpoint, along with their definitions, time each item is evaluated and the final source data for each item. Definitions provided are referenced from the Clinical Protocol, Section 3.3.

Table 1: Summary of Uncomplicated Technical Success Primary Endpoint



| Outcome | Definition (per Clinical Protocol Section 3.3) | Endpoint Time<br>Evaluated | Final Source<br>Data |
|---|---|---|---|
| Uncomplicated Technical Success | | | |
| Successful access<br>and delivery | All Gore devices are successfully tracked from the access site to the intended implantation site and released from the deliver catheter successfully without the need for unanticipated corrective intervention related to delivery. | TAMBE Device<br>Index<br>procedure | Site data |
| Successful and accurate deployment | Deployment of all required endovascular device components in the planned location: Patency of required aortic endovascular grafts with absence of device deformations (e.g., kinks) requiring unplanned placement of a non-TAMBE device component* within the endovascular graft; Patency of all branch devices with absence of device deformations (e.g., kinks) requiring unplanned placement of any non-TAMBE device component* within the branches**; * TAMBE components include the aortic component, distal bifurcated component, iliac extenders, contralateral legs, VBX component and CTAG Device. **Implantation of bare metal stents to smooth the transition from the VBX to the uncovered branch vessel will not count against technical success if the procedure otherwise meets the definition of technical success. Use of non-TAMBE devices to correct iatrogenic complications in the treated aorta or branch vessels would be considered technical failures. | TAMBE Device<br>Index<br>procedure | Site Reported<br>and CEC<br>Adjudication <sup>1</sup> |
| Successful<br>withdrawal | Successful withdrawal of the delivery systems, without a need for corrective intervention related to withdrawal | TAMBE Device<br>Index<br>procedure | Site data |
| Procedural Safety | | | |



| Outcome | Definition (per Clinical Protocol Section 3.3) | Endpoint Time<br>Evaluated | Final Source<br>Data |
|---|---|---|---|
| Aortic Rupture | Rupture in the stented segment of the aorta verified with direct observation or CT scan | 30 days | |
| Lesion-related<br>mortality | Defined as all deaths during hospitalization for index endovascular procedure and within 30 days of the index endovascular procedure or any secondary procedures due to the treated pathology, or the effectiveness of the endovascular repair (e.g., procedures to treat retrograde dissections, losses of patency, losses of device integrity, endoleaks, migrations, aortic expansions, aortic ruptures) and any deaths related to the treated pathology or endovascular graft (e.g., aneurysm rupture, retrograde dissection leading to fatal cardiac tamponade), unless evidence is available to demonstrate that the death is not lesion related | 30 days or in-<br>hospital for<br>index<br>endovascular<br>procedures | |
| Permanent<br>paraplegia | Paraplegia secondary to spinal cord ischemia identified within 30 days of the index endovascular procedure combined with spinal cord ischemia scale grade of "3" at the one-month follow-up visit. The grading system for spinal cord ischemia is described in TEVAR reporting standards | Event reported within 30 days of endovascular procedure without resolution at one month follow-up | |
| Permanent paraparesis | Paraparesis secondary to spinal cord ischemia identified within 30 days of the index endovascular procedure combined with spinal cord ischemia scale grade of "2" at the one-month follow-up visit. The grading system for spinal cord ischemia is described in TEVAR reporting standards | Event reported<br>within 30 days<br>of endovascular<br>procedure<br>without<br>resolution at<br>one month<br>follow-up | CEC<br>adjudication |
| New onset renal<br>failure requiring<br>dialysis | New onset sustained renal failure identified within 30 days of the index endovascular procedure, combined with need/requirement for dialysis at the one month follow- up visit | Event reported within 30 days of endovascular procedure without resolution at one month follow-up | |
| Severe bowel ischemia | Bowel ischemia resulting in bowel resection or fatal outcome | 30 days | |
| Disabling stroke | Stroke was assessed using the Modified Rankin Scale. Stroke identified as having occurred within 30 days of the index endovascular procedure, combined with mRS ≥2 with an increase from baseline of at least one grade at 90 days Modified Rankin Score was completed by an allied health staff member who successfully completed mRS certification or licensed medical professional | 120 days (30<br>days for Stroke<br>Events, plus 90<br>days for mRS<br>measurements) | |

<sup>1</sup>As part of successful and accurate deployment, the CEC will adjudicate use of non-TAMBE devices to correct iatrogenic complications in the treated aorta or branch vessels.

2. Clinically Significant Reintervention / Lesion Related Mortality Co-Primary Endpoint (12 months post-treatment)

**Table 2** contains the definition, endpoint time evaluated, and the final source data for the components of the Clinically Significant Reintervention / Lesion Related Mortality Co-Primary Endpoint. This endpoint is evaluated at 12 months post-treatment.

Table 2: Summary of Clinically Significant Reintervention / Lesion Related Mortality Co-Primary Endpoint

| Outcome | Definition (per Clinical Protocol Section 3.3) | Endpoint Time<br>Evaluated | Final Source Data |
|---|---|---|---|
| Clinically Significant<br>Reintervention | | | |
| Clinically-Indicated Condition | An untreated device seal zone endoleak, target-lesion growth (> 5 mm in maximum diameter) or post-treatment TAAA rupture without | 12 mo f/u visit | Core Lab (aneurysm size and endoleak) CEC Adjudication (TAAA |
| Condition | reintervention at the 12 Month window follow-up visit | | rupture) Site Data (reintervention) |
| Device Effectiveness | A compromise of a device seal zone or loss of device integrity (e.g., device kink or collapse) requiring placement of an additional stent or stent-graft | 12 mo f/u visit | |
| Subject Safety | Total occlusion of a device component, use of a bypass graft or<br>the performance of an open conversion in order to maintain bodily<br>vessel function | 12 mo f/u visit | CEC adjudication |
| Complicated Device<br>System Prophylaxis | Any device-related intervention requiring hospitalization, or extension of hospitalization, of three days or more | 12 mo f/u visit | |
| Lesion-related mortality | | | |
| Lesion-related mortality | All deaths during hospitalization for index endovascular procedure and within 30 days of the index endovascular procedure or any secondary procedures due to the treated pathology, or the effectiveness of the endovascular repair (e.g., procedures to treat retrograde dissections, losses of patency, losses of device integrity, endoleaks, migrations, aortic expansions, aortic ruptures) and any deaths related to the treated pathology or endovascular graft (e.g., aneurysm rupture, retrograde dissection leading to fatal cardiac tamponade), unless evidence is available to demonstrate that the death is not lesion related | 12 mo f/u visit | CEC adjudication |

## 2.3.2 Secondary Endpoint(s)

**Table 3** contains the definitions, endpoint time evaluated and source data for the secondary endpoints. The majority of definitions in **Table 3** are sourced from the Clinical Protocol Section 3.3. Secondary Endpoint items marked with an asterisk (\*) are defined by this document.

Table 3: Secondary Endpoint Definitions

| rabio c. Godonaary Enapoint Bonniacho | | | |
|---|---|---|---|
| Outcome | Definition | Endpoint Time Evaluated | Final Source Data |
| Standard Procedure /<br>Hospitalization Metrics | | | |
| Aneurysm-related mortality | Defined as all deaths during hospitalization for index endovascular procedure and within 30 days of the index endovascular procedure or any secondary procedures due to the treated pathology, or the effectiveness of the endovascular repair (e.g., procedures to treat retrograde dissections, losses of patency, losses of device integrity, endoleaks, migrations, | 30 Days | CEC |



| Outcome | Definition | Endpoint Time Evaluated | Final Source Data |
|---|---|---|---|
| | aortic expansions, aortic ruptures) and any deaths related to the treated pathology or endovascular graft (e.g., aneurysm rupture, retrograde dissection leading to fatal cardiac tamponade), unless evidence is available to demonstrate that the death is not lesion related. | | |
| Individual elements of Procedural Safety Aortic Rupture Lesion-related mortality Permanent paraplegia Permanent paraparesis New onset renal failure requiring dialysis Severe bowel ischemia Disabling stroke | Reference <b>Table 1</b> for definitions for these elements | Reference <b>Table 1</b> | Reference <b>Table 1</b> |
| Procedural blood loss | Estimated Blood Loss during Index Procedure (mm)* | Index Procedure | Site |
| Access-related complications | An Adverse Event determined by Site to be related to vascular access* | 30 Days | Site |
| Procedural time | Duration of Index Procedure (minutes) [the time of incision will indicate the start time and the finish time is the time of closure ]. * | Index Procedure | Site |
| Stage Procedure Time | Duration of Stage Procedure (minutes) [the time of incision will indicate the start time and the finish time is the time of closure ]. * | Stage Procedure | Site |
| Length of hospital stay | Number of Days Subject stayed in hospital (from admission date to discharge date). * | Initial Hospitalization of<br>Index Procedure | Site |
| Stage procedure length of hospital stay | Number of Days Subject stayed in hospital for<br>stage procedure (from admission date to<br>discharge date). * | Stage Procedure | Site |
| Extended Technical Clinical<br>Success | Subjects who present within the 30-Day follow-<br>up with no Type I or Type III endoleak, as<br>evaluated by CTA, and free from device-related<br>intervention | 30 Days | Core Lab |
| Aortic Stent-Graft Effectiveness<br>Measures | | | |
| Type I endoleak | Endoleak arising from the proximal or distal<br>sealing zone of a device perfusing the<br>aneurysm | Through 12 Months | Core Lab |
| Type IA endoleak | Inadequate seal at the proximal end of the device placed in the aorta | Through 12 Months | Core Lab |
| Type IB endoleak | Inadequate seal at the distal end of the device placed in iliac vessel | Through 12 Months | Core Lab |
| Type IC endoleak | Inadequate seal at the distal end of a device placed inside branch vessel | Through 12 Months | Core Lab |



| Outcome | Definition | Endpoint Time Evaluated | Final Source Data |
|---|---|---|---|
| Type II endoleak | Endoleak arising from a patent branch vessel perfusing the aneurysm, e.g., lumbar or inferior mesenteric branch | Through 12 Months | Core Lab |
| Type III endoleak | Endoleak arising from the component junction(s) of the prosthesis or due to damage to the graft material perfusing the aneurysm. | Through 12 Months | Core Lab |
| Type IIIA endoleak | Modular disconnection or apposition failure | Through 12 Months | Core Lab |
| Type IIIB endoleak | Graft tear | Through 12 Months | Core Lab |
| Type III General endoleak | A Type III endoleak whose source cannot be<br>differentiated between an intercomponent<br>junction or graft tear | Through 12 Months | Core Lab |
| Type IV endoleak | Endoleak of whole blood through the graft fabric perfusing the aneurysm | Through 12 Months | Core Lab |
| Indeterminate endoleak | Endoleak perfusing the aneurysm without a definitive source | Through 12 Months | Core Lab |
| Device Migration | Longitudinal movement of all or part of the device for a distance ≥10 mm, as confirmed by CT scan, relative to anatomical landmarks and device positioning at the first post-operative CT scan | Through 12 Months | Core Lab |
| TAAA enlargement | An increase in the maximum aneurysm diameter of 5 mm or more relative to the first post-operative CT scan within the 30 day follow-up window | Through 12 Months | Core Lab |
| Severe distal thromboembolic events | Ischemic events related to the device from tissues distal to the device implantation site sufficiently debilitating to necessitate bypass, open surgical intervention, limb amputation or leading to death | Through 12 Months | CEC |
| Aortic Rupture | Rupture in the stented segment of the aorta<br>verified with direct observation or CT Scan* | Through 12 Months | CEC |
| Device or procedure-related laparotomy | An adverse event assessed by the site as being device or procedure-related that led to a laparotomy * | Through 12 Months | Site |
| Conversion to open repair | A reintervention that resulted in explant of the device and open surgical repair* | Through 12 Months | Site |
| Aortoiliac device limb occlusion | An occlusion in the distal bifurcated component, contra-lateral limb component, contra-iliac extender component, or the ipsilateral extender component* | Through 12 Months | Core Lab |
| Loss of device integrity | Wire fracture identified in the sealing row stents of either the aortic, branch or iliac components Transient (compression) or permanent stent-graft collapse (invagination) following complete | Through 12 Months | Core Lab |

| Outcome | Definition | Endpoint Time Evaluated | Final Source Data |
|---|---|---|---|
| | device deployment, resulting in an<br>overall reduction in the aortic, branch<br>or iliac vessel luminal diameter | | |
| Primary patency<br>Adapted Study Definition | Blood flow without occlusion maintained through the device after implant without an intervention. | Through 12 Months | Site and Core Lab |
| Assisted primary patency<br>Adapted Study Definition | Blood flow maintained through the device after implant regardless of re-interventions performed (without occlusion) | Through 12 Months | Site and Core Lab |
| Secondary patency<br>Adapted Study Definition | Blood flow through the device regardless of<br>reinterventions performed (with or without<br>occlusion) and freedom from surgical bypass | Through 12 Months | Site and Core Lab |
| All reinterventions | An additional unanticipated interventional or surgical procedure (including conversion to open surgery), related to the device (including withdrawal of the delivery system) or procedure. Anticipated or unanticipated status will be determined at the discretion of the investigator. | Through 12 Months | Site |
| | These will not include unanticipated, corrective intervention at the access site(s), or device intervention to address non-treatment area issues | | |
| Branch Vessel Device<br>Effectiveness Measures | | | |
| Branch vessel patency | Primary, Assisted Primary, Secondary Patency | 12 Months | Site and Core Lab |
| Acute kidney injury | >50% decrease in eGFR within 30 days of TAMBE Device treatment when compared to pre-treatment serum creatinine value | 30 days | Site |
| Renal function deterioration | A sustained >25% decrease in eGFR over two consecutive study visits following TAMBE Device treatment when compared to pretreatment serum creatinine value | 12 Months | Site |

## 2.4 Statistical Hypotheses

The analysis of the Uncomplicated Technical Success / Procedural Safety endpoint is intended to test the hypothesis that the safety of the TAMBE Device exceeds the performance goal of 80% technical success. This analysis will be performed on the Primary Study Arm (pararenal aortic aneurysms and adapted Crawford Type IV TAAA). The analysis of the Clinically Significant Reintervention / Lesion Related Mortality endpoint is intended to test the hypothesis that the effectiveness of the TAMBE Device exceeds the performance goal of 68% free from clinically significant reintervention / lesion related mortality events.

The hypotheses are specified as follows:

<u>Uncomplicated Technical Success / Procedural Safety Hypothesis:</u>



$$H_0: P_{UCT} \le 0.80$$

$$H_A: P_{UCT} > 0.80$$

Where  $P_{UCT}$  denotes the proportion of subjects that achieve technical success.

# Clinically Significant Reintervention / Lesion Related Mortality Hypothesis:

$$H_0: P_{CSR} \leq 0.68$$

$$H_A: P_{CSR} > 0.68$$

Where  $P_{CSR}$  denotes the proportion of subjects that achieve freedom from clinically significant reintervention.

2.5



#### 2.6 Sample Size Calculations

Sample size calculations were determined using PASS 13.0.8 ("Tests for One Proportion using Proportions" and "Exact" options).

The sample size calculation was motivated primarily by the Clinically Significant Reintervention Hypothesis / Lesion Related Mortality, since that would require more subjects to properly power than the Uncomplicated Technical Success / Procedural Safety hypothesis.

At least 86 are required to maintain > 80% power for the Clinically Significant Reintervention / Lesion Related Mortality Hypothesis. Assuming a 15% loss-to-follow-up rate, 102 subjects are sufficient for achieving the objective (with 81.48% power). For uncomplicated technical success, a sample size of 102 enrolled and implanted subjects (86 expected evaluable subjects) will yield a power of 93.41%. We expect the results of these hypotheses tests to be correlated, so an overall power calculation of the product of the two powers is inappropriate.

Expected accrual of subjects for the Primary Study Arm is 27 to 32 months.

# 3. Study Treatment Arms

## 3.1 Test Arms

There will be a Primary Study Arm and a Secondary Study Arm in this study.

- Primary Study Arm Hypothesis-driven analysis, TAAAs which are anatomically suitable for treatment with the TAMBE System and do not require proximal extension with a CTAG Device (N=102)
- Secondary Study Arm Non hypothesis-driven analysis, TAAAs which are anatomically suitable for treatment with the TAMBE System and would require proximal extension with CTAG Device(s) (N=20 minimum,100 maximum as aggregate total of all types). Subjects that undergo placement of the CTAG Device but do not complete the implant of the TAMBE Device whether by subject choice or Investigator discretion will only have their adverse events reported through 30 days after implant and withdrawn from the study.

## 3.2 Control Arm(s)

There are no control arms in this study.

## 4. Study Data Collection

Subjects will be evaluated, at a minimum, using the schedule of events described in **Table 4**. The timing of study evaluations will be done according to the schedule defined in **Table 5**. Investigators will be held responsible for the performance of all Protocol-required testing at their respective time points, including testing done at institutions different than the implanting study site. It is highly recommended that subjects return back to their centers of enrollment for follow-up evaluations to foster testing compliance and continuity of care.

Sites are to schedule all study testing to be performed within the ideal visit window; however, any available data collected in the analysis window will be summarized as occurring within the given window. Data collected outside the ideal window, but within the analysis window will not be considered a protocol deviation.

#### 4.1 Study Collection Intervals

Subjects will be asked to return for follow-up visits at one (1), three (3), six (6), 12, 24, 36, 48, and 60 months post-treatment. At each follow-up visit, subjects will undergo an evaluation for adverse events.

| | Pre-<br>treatment<br>(Screening) | Treatment | Hospital<br>Discharge | One<br>Month | Three<br>Months | Six<br>Months | Annually through 5 Years |
|---|---|---|---|---|---|---|---|
| Informed Consent | X | | | | | | |
| Demographics and<br>Medical History | Х | | | | | | |
| Risk Scales<br>(ASA, NYHA, SVS) | Х | | | | | | |
| Physical examination | X | × 83 | X | X | X | X | X |
| Adverse Events | X | X | X | X | X | X | X |
| Medication<br>Review | Х | | X | Х | Х | X | Х |
| Modified Rankin<br>Scale <sup>a,b</sup> | X | | X | х | X<br>If<br>applicable | Х | |
| Spinal Cord Ischemia Scale <sup>a</sup> | Х | 30 | Х | Х | | Х | |

Table 4: Schedule of Events



| NIH Stroke Scale <sup>c</sup> | Х | | X<br>If<br>applicable | | | | |
|---|---|---|---|---|---|---|---|
| SF-36 Questionnaire | X | | | X | X | X | X |
| Serum Creatinine<br>Concentration | Х | | Х | X | Х | Х | Х |
| Spiral CTA (contrast) | X | | | X | | Х | X |
| Spiral CT (non-<br>contrast) | | | | Х | | X<br>Optional | X<br>Optional |
| Completion<br>Angiogram | | Х | | | | | VI. |
| Magnified Branch<br>Visualization | | X | | | | | |
| Abdominal<br>Ultrasound | X | | Х | X | X | х | Χ |
| Multiplanar Device<br>Radiographs (X Ray) | | | | Х | | х | Х |

<sup>&</sup>lt;sup>a</sup> If subject is unable to return to the site for a follow-up visit, they may be contacted by telephone to evaluate the Modified Rankin Scale and Spinal Cord Ischemia Scale.

<sup>&</sup>lt;sup>b</sup> For subjects suspected of having a stroke event within 30 days following the index endovascular procedure an additional mRS score should be completed at 90 days following the suspected stroke event but no greater than 120 days post index endovascular procedure.

c NIH Stroke Scale should be performed for any subject suspected of having a stroke event that undergoes the treating site's stroke protocol during the study interval from the initiation of the index endovascular procedure until discharge. The scale should be performed as soon as possible after learning of the suspected event and again at the time of discharge.

possible after learning of the suspected event and again at the time of discharge.

d CTA of chest/abdomen/pelvis at Screening. CTA of abdomen and pelvis at all follow-up visits, except for Secondary Study Arm Subjects who must have a CTA of chest/abdomen/pelvis at all visits. MRA may be used in place of CTA during follow-up if the Subject is contraindicated for CTA.

# 4.2 Follow-up Visit Windows

Follow-up visits will be scheduled at appointed times after the date of treatment. The Sponsor recognizes that Subjects may not be able to return for follow-up visits on the exact date required. Thus, a period during which each visit is allowed is demonstrated in **Table 5**.

Table 5: Follow-up Visit Ideal and Analysis Window Definitions

| Follow-up Visit | Ideal Window (days) | Analysis Window (days) |
|-----------------|---------------------------|------------------------|
| Procedure | 0 | 0 |
| Discharge* | Before hospital discharge | N / A |
| Post-Procedure | Not required | 1-14 |
| 1 Month | 23-44 | 15-59 |
| 3 Month | 76-104 | 60-126 |
| 6 Months | 150-210 | 127-242 |
| 12 Months | 275-455 | 243-546 |
| 24 Months | 640-820 | 547-911 |
| 36 Months | 1005-1185 | 912-1275 |
| 48 Months | 1370-1550 | 1276-1640 |
| 60 Months | 1735-1915 | 1641-2006 |

<sup>\*</sup>Follow-up visit is categorized as "Discharge" through initial hospitalization, regardless of length.

#### 4.3 Data and Safety Monitoring Board

See Section 9.3 of the protocol for information on the Data and Safety Monitoring Board.

#### 4.4 Clinical Event Committee

See Section 9.4 of the protocol for information on the Clinical Events Committee.

## 4.5 Site Enrollment Restrictions

The maximum number of implanted subjects that may be implanted at a single site is as follows:

- Primary Study Arm Subjects: 15 subjects
  - Continued Access + Primary Study Arm: 21 subjects (this is a temporary site maximum which will be lifted after the first 27 subjects have enrolled in Continued Access)
- Secondary Study Arm Subjects: No maximum

#### 4.6 Core Lab

See Section 6.4 of the protocol for information on the Core Lab.

#### 4.7 Handling of Missing Dates

Imputation of dates is not planned for Primary Analysis. However, if it becomes necessary for an analysis of adverse events, the earliest possible date will be used, given the information available. If the month and year are provided, but the day is missing, then the first day of the month will be imputed. If only the year is provided, then the first day of the first month will be imputed, or the first day after procedure imputed if the first day of the year is prior to the procedure.

## 5. Statistical Analyses

#### 5.1 Analysis Populations

The following populations will be used in various analyses of the data collected in the AAA 17-01 study:

- All Enrolled Subjects This population will consist of all enrolled Subjects. A patient is considered enrolled into the study once the Main informed consent has been signed and dated.
- All Enrolled and Implanted Subjects This population will consist of all enrolled and implanted Subjects. A patient is considered enrolled into the study once the Main informed consent has been signed and dated, and successfully implanted with the study device (TAMBE in the primary arm, CTAG + TAMBE in the secondary arm).
- 3. Uncomplicated Technical Success Eligible Population (each study arm) [Per protocol population] This population will consist of enrolled and implanted Subjects with a follow-up visit at or after 30 days following initial TAMBE Device implant procedure. Additionally, any Subjects with an eligible technical success event, as defined in Section 2.3.1, even if they did not complete a follow-up visit at or after 30 days following initial procedure, will be included.
- 4. <u>Clinically Significant Reintervention / Lesion Related Mortality Population (each study arm)</u> This population will consist of enrolled and implanted Subjects that have completed the 12 month analysis window. Additionally, any Subjects with an eligible clinically significant reintervention event, as defined in **Section 2.3.1**, even if they did not complete the necessary follow-up visit or imaging to otherwise be included in the population, will be included.
- Secondary Effectiveness Populations (each study arm, each endpoint) These
  populations will consist of enrolled Subjects with an evaluable result for the specific
  variable.
- Reduced Profile VBX Population This population will consist of the subjects in the Continued Access Phase who had been implanted with at least one reduced profile VBX device.

#### 5.2 Endpoint Variables

The sources for the endpoint variables can be found in **Table 1**, **Table 2**, and **Table 3** in **Section 2.3.1** and **Section 2.3.2**.

#### 5.3 Timing of Analyses

The Uncomplicated Technical Success / Procedural Safety endpoint will be analyzed after all Subjects eligible for the Primary Arm Uncomplicated Technical Success / Procedural Safety Eligible Population have completed a follow-up visit in the 12 month follow-up window and have been on the study for 90 days.

The Clinically Significant Reintervention endpoint will be analyzed after all Subjects eligible for the Primary Arm Clinically Significant Reintervention Eligible Population have completed a follow-up visit in the 12 month window.

The primary safety endpoint will be analyzed in the Primary Study arm during the effectiveness analysis.



The Primary and Secondary Study arms will be treated independently from each other, with the secondary study arm limited to descriptive analysis.

The Sponsor will collect data that comprise the secondary endpoints throughout all study follow-up (5 years), as appropriate, in addition to their specified analysis times (see **Section 4.2**). For endpoint events that rely on CEC adjudication, site reported data will be used to assess endpoints after the 12 month analysis period.

Following accrual of the initial 102 study subjects into the Core Clinical Investigation, up to 65 additional study subjects will be enrolled and implanted to allow for Continued Access to the device after the original enrollment is complete. The initial and additional subjects will be evaluated per the Inclusion / Exclusion criteria and will employ the same follow-up schedule. All statistical inference for the PMA submission will be based on the initial 102 subjects. Data from subjects enrolled in the Continued Access cohort will be reported separately but may be pooled with the initial data for subsequent follow-up reports.

Analyses of the reduced profile VBX Device will be completed once a minimum of 10 subjects (of the Continued Access phase) are enrolled and implanted with reduced profile VBX Device and followed through 30 days

#### 5.4 Statistical Analysis of Endpoints

One-sided exact Clopper-Pearson confidence intervals for binomial proportions (alpha=0.05) will be constructed to test the Uncomplicated Technical Success and Clinically Significant Reintervention hypotheses in the Primary Study Arm. The null hypothesis for each endpoint will be rejected if the lower bounds of the 95% confidence interval exceeds the corresponding performance goal. This is equivalent to stating that the estimated effectiveness and safety must exceed the PG with a Type I error rate (alpha) of < 0.05.

Primary and Secondary Endpoints will be summarized in the Secondary Study Arm, but no hypotheses tests will be performed.

All events must meet the protocol definition.

#### 5.4.1 Uncomplicated Technical Success / Procedural Safety Endpoint Events

Uncomplicated Technical Success endpoint events in each study arm will be computed as all enrolled Subjects experiencing an event meeting the definition in **Section 2.3.1.** 

5.4.2 Clinically Significant Reintervention / Lesion Related Mortality Events Endpoint Events

Clinically Significant Reintervention endpoint events in each study arm will consist of all enrolled Subjects experiencing an event meeting the definition in **Section 2.3.1**.

#### 5.5 Adverse Events

The definition for Anticipated Adverse Events is given in Section 9.1 of the protocol. Section 9.1.1 describes the assessment of AE relationships, Section 9.1.2 describes determination of seriousness, and Section 9.1.3 describes their reporting and coding.











# 6. Interim Analyses and Safety Monitoring Analyses (if applicable)

Safety data will be periodically reviewed by a Data Safety and Monitoring Board (DSMB), but these reviews will not constitute statistical analyses and therefore no adjustments for multiple testing will be necessitated. A comprehensive summary of all reported adverse events will be reviewed.

# 7. Analysis Specifications



## 7.3 Verification Level for Statistical Output

All necessary analysis datasets as well as tables referenced herein will be verified at Level I. All listings referenced herein will be verified at Level II. Verification levels are explained in MD111325 Clinical Affairs Biostatistics Analysis Specification and Programming.

# 8. Data Sets, Tables, Figures, and Listings

This section includes a list of the minimal planned statistical outputs, including tables, listings and figures which are to be created for the regulatory reports defined in the protocol. A different selection of tables, listings, and figures can be created for all other reporting efforts (DSMB, Annual Report, etc.) as decided necessary. Dataset names and descriptions may also be included.





9.